CLINICAL TRIAL: NCT01332266
Title: An Open-Label, Multicenter, Randomized, Phase 1b/2 Study of E7050 in Combination With Cetuximab Versus Cetuximab Alone in the Treatment of Platinum-Resistant Squamous Cell Carcinoma of the Head and Neck
Brief Title: E7050 in Combination With Cetuximab Versus Cetuximab Alone in the Treatment of Platinum-Resistant Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PharmaBio Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7050-702; 2011-000773-31 (EudraCT Number)
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2017-12

CONDITIONS: Platinum-Resistant Squamous Cell Carcinoma of the Head and Neck
Keywords: Cancer; head and neck; squamous cell carcinoma of the head and neck; phase 1b; phase 2
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Active Comparator; Phase 1b: Cohort 1,2,and 3 (Active Comparator): Phase 1b:
  Cohort 1; 200 mg E7050 + 250 mg/m2 cetuximab Cohort 2; 300 mg E7050 + 250 mg/m2 cetuximab Cohort 3; 400mg E7050 + 250mg/m2 cetuximab
  Phase 2: Arm 1; MTD E7050 + 250 mg cetuximab Arm 2; 250 mg cetuximab
  Interventions: Drug cetuximab
  Interventions: Drug: E7050; Drug: Cetuximab
- Phase 2 (Active Comparator): Phase 2:
  Arm 1; MTD E7050 + 250 mg/m2 cetuximab Arm 2; 250 mg/m2 cetuximab
  Interventions: Drug: E7050; Drug: Cetuximab

INTERVENTIONS:
Drug: E7050 — E7050 given orally at 200, 300, or 400 mg once daily.
  Other Names: Golvatinib
Drug: Cetuximab — Cetuximab is given at an initial dose of 400 mg/m2 given as a 2-hour intravenous (IV) infusion on Day 1 of Cycle 1, followed by a dose of 250 mg/m2 given as a 1-hour IV infusion on Day 8, Day 15, and Day 22 of Cycle 1, and Day 1, Day 8, Day 15, and Day 22 of each subsequent cycle.

SUMMARY:
The purpose of this study is to determine whether participants with platinum-resistant squamous cell carcinoma of the head and neck (SCCHN) who receive either E7050 administered with cetuximab or cetuximab alone experience greater benefit.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of a Phase 1b: a safety run-in period with 3 ascending doses of E7050 in combination with cetuximab; and a Phase 2 portion: a randomized 2-arm period. Approximately 95 participants with platinum-resistant squamous cell carcinoma of the head and neck will be enrolled in the study (10-15 participants in the Phase 1b portion and 80 participants in the Phase 2 portion). Participants will only participate in either the Phase 1b or the Phase 2 portion of the study.

In the Phase 2 portion, participants will receive study treatment (E7050 plus cetuximab or cetuximab alone) for approximately six 28-day cycles (24 weeks). Beyond 24 weeks, participants who are experiencing clinical benefit may continue E7050 plus cetuximab, cetuximab alone or E7050 alone (Arm 1), or may continue cetuximab alone (Arm 2), depending on the original randomization treatment arm, for as long as clinical benefit is sustained and the treatment is well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Platinum-resistant (defined as failure to respond to treatment with a platinum agent or recurrence of disease after initial response to platinum within 12 months of completing therapy), locally advanced, recurrent and/or metastatic SCCHN, which is untreatable by surgical resection or radiation therapy
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* Blood pressure must be well-controlled. Participants must have no history of hypertensive crisis or hypertensive encephalopathy; Adequate end organ function

Exclusion Criteria

* Nasopharyngeal tumors
* Previously received E7050, anti-angiogenic therapy, or anti-epidermal growth factor receptor (EGFR) therapy (prior anti-angiogenic/EGFR therapy is permitted in Phase 1b only. Prior cetuximab is permitted if administered in combination with radiation
* Presence of brain metastases, unless the participant has received adequate treatment at least 4 weeks prior to randomization, and is stable, asymptomatic, and off steroids for at least 4 weeks prior to randomization
* Palliative radiotherapy is not permitted throughout the study period
* Clinically significant hemoptysis
* Serious non-healing wound, ulcer, or active bone fracture
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1, or anticipation of need for a major surgical procedure during the course of the study
* Clinically significant gastrointestinal bleeding within 6 months prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2017-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (7):
  - Tucson, Arizona
  - Fort Myers, Florida
  - Boston, Massachusetts
  - St Louis, Missouri
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
- South Korea (4):
  - Goyang-si, Gyeonggi-do
  - Hwasun, Jeollanam-do
  - Busan
  - Seoul
- Ukraine (5):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Sumy
- United Kingdom (3):
  - London, Greater London
  - Manchester, Greater Manchester
  - Glasgow, Strathclyde

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 28 investigative sites in the Republic of Korea, Ukraine, United Kingdom, and the United States from 19 September 2011 to 04 September 2017.
Pre-assignment Details: This study consists of two phases Phase 1b and Phase 2. Phase 1b: 12 participants were enrolled and received the study treatment; Phase 2: 83 participants were enrolled and received the study treatment.
Groups:
- Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant squamous cell carcinoma of the head and neck (SCCHN) received golvatinib 200 milligram (mg) tablets, orally, once daily (run-in period) and cetuximab 400 milligram per square meter (mg/m^2) intravenous infusion, once on Day 1 of Cycle 1, followed by cetuximab 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles for determining maximum tolerated dose (MTD) or Recommended Phase 2 dose (RP2D), until the occurrence of progressive disease (PD), unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received golvatinib 300 mg tablets, orally, once daily (run-in period) and cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by cetuximab 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles for determining MTD or RP2D, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received golvatinib 400 mg tablets, orally, once daily (run-in period) and cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by cetuximab 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles for determining MTD or RP2D, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received golvatinib 400 mg (RP2D) tablets, orally, once daily and cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by cetuximab 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles. After 6 cycles, at the discretion of the investigator, participants who experienced clinical benefit could continue for as long as clinical benefit was sustained and the treatment was well tolerated, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 2: Arm 2: Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles. After 6 cycles, at the discretion of the Investigator, participants who experienced clinical benefit could continue for as long as clinical benefit was sustained and the treatment was well tolerated, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Period: Phase 1b
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Started | 4 | 5 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 5 | 3 | 0 | 0
Not completed — Death | 3 | 3 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Started | 0 | 0 | 0 | 42 | 41
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 42 | 41
Not completed — Death | 0 | 0 | 0 | 33 | 36
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 3 | 1
Not completed — Symptomatic deterioration | 0 | 0 | 0 | 0 | 1
Not completed — Progression Disease | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants enrolled and randomized into Phase 1b and Phase 2, except for those who drop out of study prior to receiving any study treatment, or were without any safety assessments following the first dose of study treatment.
Groups:
- Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received golvatinib 200 mg tablets, orally, once daily (run-in period) and cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by cetuximab 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles for determining MTD or RP2D, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2 | Total
Number analyzed (Participants) | 4 | 5 | 3 | 42 | 41 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (8.29) | 58.8 (12.58) | 59.3 (5.51) | 58.4 (11.04) | 53.9 (9.84) | 57.0 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 4 | 7 | 13
  Male | 2 | 5 | 3 | 38 | 34 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 5 | 3 | 41 | 41 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 3 | 16 | 12 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 2
  White | 2 | 1 | 0 | 24 | 29 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0=Fully Active (Most Favorable Activity); 1=Restricted activity but ambulatory; 2=Ambulatory but unable to carry out work activities; 3=Limited Self-Care; 4=Completely Disabled, No self-care (Least Favorable Activity); 5=Dead.
  Participants
    ECOG: 0 (Fully Active) | 1 | 0 | 0 | 10 | 10 | 21
    ECOG: 1 (Restricted in Physical Activity; Ambulatory) | 3 | 4 | 3 | 28 | 24 | 62
    ECOG: 2 (Ambulatory and Capable of All Self-care) | 0 | 1 | 0 | 1 | 3 | 5
    ECOG: 3 (Capable of Only Limited Self-care) | 0 | 0 | 0 | 0 | 0 | 0
    ECOG: 4 (Completely Disabled) | 0 | 0 | 0 | 0 | 0 | 0
    ECOG: 5 (Dead) | 0 | 0 | 0 | 0 | 0 | 0
    Not Specified | 0 | 0 | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-limiting Toxicities (DLTs) as Per National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0)
Description: DLT:adverse events graded as NCI CTCAEv4.0 occurring less than or equal to(<=)28 days after treatment.Events as: Non-hematological: 1)Grade greater than or equal to(>=)3 peripheral neuropathy; 2)Grade 3 fatigue or 2 point decline in eastern cooperative oncology group performance status that persisted for greater than(>)7 days; 3)Grade >=3 nausea,vomiting despite optimal antiemetic treatment; 4)Any nonhematologic toxicity of Grade >=3, with exceptions as alopecia,single laboratory values out of normal range,hypersensitivity reaction. Hematological 1)Grade 4 neutropenia lasting >7 days; 2)Febrile neutropenia as fever >=38.5 degree celsius with absolute neutrophil count less than(<)1.0*10^9 per liter(/L); 3)Grade 3 thrombocytopenia with nontraumatic bleeding requiring platelet transfusion; 4)Grade 4 thrombocytopenia with/without nontraumatic bleeding. Other 1)Study drug related death; 2)Toxicity that dose escalation committee believed to be DLT that was not covered by above DLT criteria.
Time Frame: Cycle 1 (Cycle length is equal to [=] 28 days)
Population: Safety population was defined as all participants enrolled and randomized to treatment in study, except for those who drop out of the study prior to receiving any study treatment, or were without any safety assessments following the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received 200 mg of golvatinib tablets orally, once daily (run-in period) and Cetuximab 400 mg/m^2 as intravenous infusion, once on day 1 of cycle 1, followed by 250 mg/m^2 as intravenous infusion, once on days 8, 15 and 22 of cycle 1 of 28-days treatment cycle for 6 subsequent cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received 300 mg of golvatinib tablets orally, once daily (run-in period) and Cetuximab 400 mg/m^2 as intravenous infusion, once on day 1 of cycle 1, followed by 250 mg/m^2 as intravenous infusion, once on days 8, 15 and 22 of cycle 1 of 28-days treatment cycle for 6 subsequent cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
- Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2: Participants with platinum-resistant SCCHN received 400 mg of golvatinib tablets orally, once daily (run-in period) and Cetuximab 400 mg/m^2 as intravenous infusion, once on day 1 of cycle 1, followed by 250 mg/m^2 as intravenous infusion, once on days 8, 15 and 22 of cycle 1 of 28-days treatment cycle for 6 subsequent cycles until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 4 | 5 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Phase 1b: Plasma Concentration of Golvatinib When Given in Combination With Cetuximab
Time Frame: Cycle 1: 0-48 hours post-dose (Each cycle=28 days)
Population: Data was not collected and analyzed for this outcome measure because no pharmacokinetic analysis was conducted in this study due to incomplete pharmacokinetic sample bioanalysis due to unresolved queries leading to inadequate calculations and limited data interpretability.
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Phase 2: Number of Participants With Grade 3 or Higher Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as an adverse event that has an onset date, or a worsening in severity from baseline (pre-golvatinib), on or after the first dose of golvatinib. The severity was graded according to CTCAE v4.0. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to adverse event.
Time Frame: Up to 5 years 11 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
Participants | 21 | 21

4. Primary Outcome: Phase 2: Number of Participants With Markedly Abnormal Vital Sign Values
Time Frame: Up to 4 years 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
Participants | 0 | 0

5. Primary Outcome: Phase 2: Number of Participants With Markedly Abnormal Physical Examinations Findings
Description: Physical examination was performed and included evaluation of 1) General appearance, 2) Head; Eyes; Ears; Nose; Throat (HEENT), 3) Neck, 4) Heart, 5) Chest (Including Lungs), 6) Abdomen, 7) Extremities, 8) Skin, 9) Lymph Nodes, and 10) neurological status. Here, number of participants with markedly abnormal physical examinations were reported.
Time Frame: Up to 4 years 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
Participants
  General Appearance | 5 | 6
  HEENT | 20 | 17
  Neck | 24 | 22
  Heart | 1 | 0
  Chest (Including Lungs) | 4 | 5
  Abdomen | 6 | 3
  Extremities | 2 | 0
  Skin | 4 | 5
  Lymph Nodes | 13 | 15
  Neurologic | 3 | 5

6. Primary Outcome: Phase 2: Number of Participants With Markedly Abnormal Electrocardiogram (ECG) Values
Time Frame: Up to 4 years 4 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
Participants | 0 | 0

7. Secondary Outcome: Phase 2: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of randomization until the earlier of the following two events: the date of PD or the date of death based on response evaluation criteria in solid tumor (RECIST) v1.1. PD is defined as at least a 20 percent (%) increase or 5 millimeter (mm) increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS was estimated and analyzed using Kaplan Meier method. As planned, data for this endpoint was analyzed and collected till primary completion date.
Time Frame: From the date of randomization until the earlier of the following two events: the date of PD or the date of death (Up to approximately 4 years 4 months)
Population: Modified Intent-to-Treat (MITT) analysis set included all participants randomized in the applicable study arm who received any comparator or study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
weeks | 15.71 [12.14 to 23.86] | 15.71 [9.29 to 18.71]
Statistical Analysis 1: Comparison: Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 vs Phase 2: Arm 2: Cetuximab 400 mg/m^2; Test type: Superiority; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.54 to 1.46]

8. Secondary Outcome: Phase 2: Percentage of Participants With PFS at Week 12
Description: PFS rate at week 12 is defined as the percentage of participants who were still alive without disease progression at 12 weeks from the date of randomization. PFS is defined as the time from the date of randomization until the earlier of the following two events: the date of PD or the date of death based on RECIST v1.1. PD is defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. PFS rate was estimated and analyzed using Kaplan Meier method.
Time Frame: At Week 12
Population: MITT analysis set included all participants randomized in the applicable study arm who received any comparator or study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
percentage of participants | 68.9 [50.79 to 81.44] | 59.4 [41.90 to 73.23]

9. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization until the date of PD based on RECIST v1.1. PD is defined as at least a 20% increase or 5 mm increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) recorded since the treatment started or the appearance of 1 or more new lesions. TTP was estimated and analyzed using Kaplan Meier method. As planned, data for this endpoint was analyzed and collected till primary completion date.
Time Frame: From the date of randomization until the date of PD (Up to approximately 4 years 4 months)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
weeks | 15.43 [12.14 to 23.14] | 16.00 [9.29 to 19.14]
Statistical Analysis 1: Comparison: Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 vs Phase 2: Arm 2: Cetuximab 400 mg/m^2; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.61 to 1.73]

10. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until the date of death. OS was analyzed using Kaplan Meier method. As planned, data for this endpoint was analyzed and collected till primary completion date.
Time Frame: From the date of randomization until the date of death (Up to approximately 4 years 4 months)
Population: MITT analysis set included all participants randomized in the applicable study arm who received any comparator or study drug. Here "Overall number of participants analyzed" signifies participants with events (death).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 33 | 36
weeks | 39.71 [28.43 to 49.71] | 36.71 [28.00 to 44.43]
Statistical Analysis 1: Comparison: Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 vs Phase 2: Arm 2: Cetuximab 400 mg/m^2; Test type: Superiority; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.53 to 1.37]

11. Secondary Outcome: Phase 2: Percentage of Participants With Overall Response
Description: Overall response rate is defined as percentage of participants with complete response (CR) or partial response (PR) based on RECIST v1.1. CR is defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As planned, data for this endpoint was analyzed and collected till primary completion date.
Time Frame: From the date of randomization until CR or PR (Up to approximately 4 years 4 months)
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2: Arm 2: Cetuximab 400 mg/m^2: Participants with platinum-resistant squamous cell carcinoma of the head and neck received cetuximab 400 mg/m^2 intravenous infusion, once on Day 1 of Cycle 1, followed by 250 mg/m^2 intravenous infusion, once on Days 8, 15 and 22 of Cycle 1 in a 28-days treatment cycle for up to 6 subsequent cycles. After six cycles, at the discretion of the Investigator, participants experienced clinical benefit have continued for as long as clinical benefit was sustained and the treatment was well tolerated, until the occurrence of PD, unacceptable toxicity, withdrawal of consent, withdrawal by the Investigator, lost to follow-up, or death, whichever occurred first.
Arm/Group | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
Number analyzed (Participants) | 42 | 41
percentage of participants | 9.5 [0.7 to 18.4] | 4.9 [0 to 11.5]

ADVERSE EVENTS:
Time Frame: Up to 5 years 11 months
Arm/Group | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 | Phase 2: Arm 2: Cetuximab 400 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/5 | 2/3 | 33/42 | 36/41
Serious Adverse Events (participants affected / at risk) | 1/4 | 4/5 | 2/3 | 15/42 | 15/41
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 3/3 | 42/42 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 (N=4) | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 (N=5) | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 (N=3) | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 (N=42) | Phase 2: Arm 2: Cetuximab 400 mg/m^2 (N=41)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Upper Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mechanical Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Cavity Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1: Golvatinib 200 mg + Cetuximab 400 mg/m^2 (N=4) | Phase 1b: Cohort 2: Golvatinib 300 mg + Cetuximab 400 mg/m^2 (N=5) | Phase 1b: Cohort 3: Golvatinib 400 mg + Cetuximab 400 mg/m^2 (N=3) | Phase 2: Arm 1: Golvatinib 400 mg + Cetuximab 400 mg/m^2 (N=42) | Phase 2: Arm 2: Cetuximab 400 mg/m^2 (N=41)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (8) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (9) | 10 (12) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 19 (35) | 3 (3)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 3 (4) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 1 (1) | 0 (0) | 4 (5) | 5 (6)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 1 (1) | 2 (2) | 10 (13) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 10 (22) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (6) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (3) | 2 (2) | 10 (10) | 2 (3)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 10 (12) | 3 (3)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 2 (3) | 10 (17) | 7 (9)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1) | 2 (3) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (6) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 4 (10) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein Total Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 19 (22) | 8 (9)
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (12)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eastern Cooperative Oncology Group Performance Status Worsened (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 14 (19) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
No pharmacokinetic analysis was conducted in this study due to incomplete pharmacokinetic sample bioanalysis due to unresolved queries leading to inadequate calculations and limited data interpretability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes